CLINICAL TRIAL: NCT00769262
Title: Effect of Conservative Weaning of Thermoregulatory Support on Weight Gain and Length of Stay in Preterm Neonates
Brief Title: Weaning Thermoregulatory Support in Preterm Neonates
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient resources to conduct study
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1105137
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Premature Neonates
Keywords: Premature neonates; Thermoregulation; Isolette; Feeding status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aggressive Weaning (Active Comparator): Infants will be weaned from the isolette using our current NICU standard of care.
  Interventions: Other: Aggressive Weaning
- Conservative Weaning (Experimental): Infants will be weaned from the isolette using a modified conservative weaning schedule.
  Interventions: Other: Conservative weaning

INTERVENTIONS:
Other: Conservative weaning — Infants will not be weaned from the isolette until their feeds are at full calorie goal (120 kcal/kg/day) and at least half of feeds are taken orally.
  Arms: Conservative Weaning
Other: Aggressive Weaning — Infants will be weaned from the isolette based solely on their temperature without regard to feed status (current standard of care in our NICU)
  Arms: Aggressive Weaning

SUMMARY:
Preterm newborns typically must be thermally regulated. In the United States, isolettes (incubators) are used to help them maintain their temperature. Traditionally, the temperature support (i.e. the temperature of the incubator) is decreased slowly according to NICU protocol until the baby is able to maintain its temperature in an open crib, without regard to the status of its feedings. This study will attempt to determine if there is a difference in length of stay, weight gain, and calories needed to gain appropriate weight between a group of newborns whose isolette temperatures are decreased in an aggressive strategy (isolette temperatures are decreased based only on baby's body temperature), and a group of newborns whose isolette temperatures are decreased in a conservative strategy (isolette temperatures are decreased to a minimum temperature and then kept steady until their feeds are at caloric goal and they are taking at least half of their feeds by mouth).

DETAILED DESCRIPTION:
General Background:

There are three key milestones premature infants must meet prior to discharge from the NICU:

1. The ability to maintain their temperature in an open crib
2. The ability to consume enough calories for adequate growth by oral feeds
3. A demonstrated weight gain consuming these feeds.

It is well understood that infants must increase their resting metabolic rate when weaned from the isolette to an open crib (1, 6). Preterm neonates have less metabolic reserve (brown fat) to allow them to mount an appropriate thermogenic response to cold stress (4). The reserve they do have is often depleted at delivery, leaving them with little or no reserve (4). When a neonate is challenged to maintain its body temperature, it must increase heat production which may affect weight gain (3). Some institutions wean without regard to neonate's weight or feeding status, while others only begin the weaning process at a predetermined weight. Currently neonates are weaned from their isolettes based largely on the traditions and experiences of clinicians, without regard to their feeding status. However, there is currently very little evidence in the literature to inform practice on the ideal conditions for weaning a neonate from their isolette. An extensive literature review has revealed no published data regarding the relationship of feed status to success at isolette weaning.

The transfer to open crib is important; if the neonate is not able to maintain his/her temperature, the length of stay could be lengthened and weight gain adversely affected (3). Cold stress can also cause adverse clinical effects including lethargy, hypotonia, poor feeding, abdominal distention, vomiting, pallor, tachypnea, and respiratory distress (2). These adverse clinical effects may also lengthen cost and length of stay, as well as adversely affect feeding. Furthermore, a return to the isolette can be quite stressful to parents and family members (3).

Subjects:

Approximately 110 subjects will be recruited. The subjects for this study will be live born preterm infants between 26 and 0/7 weeks gestation and 34 and 6/7 weeks gestation. Informed consent will be obtained from the parents.

Methods:

Neonates will be randomly assigned to either the control group (with standard thermoregulatory weaning protocol) vs. experimental group (with conservative thermoregulatory weaning protocol). After an infant is enrolled in the study, an envelope indicating random assignment to either the aggressive or conservative group will be drawn and the infant will be assigned to the indicated study group. The envelopes will be provided by the statistician and will be delivered in groups of 10 to ensure relatively equal numbers of babies in both study groups.

All infants will be advanced to goal caloric feeds of 120 Kcal/kg. Weight gain will be measured biweekly, and if adequate weight gain (average 20 grams/kg/day) is not reached, feeds will be advanced by 10 Kcal/kg/day biweekly until adequate weight gain is reached.

All infants will be kept on skin control mode until they weigh 1500 grams. Babies on skin control mode will be unclothed except for a diaper. Once infants reach 1500 grams, they will be placed on air control mode. Babies on air control mode will be dressed in one medium-weight sleeper with feet (or with socks if sleeper is footless), one hat, and no blankets or other clothing.

Control Group: Aggressive Wean

Weaning Process:

* If baby's temperature is greater than or equal to 36.7°C on 2 consecutive measurements 3 hours apart, the isolette set temperature will be lowered by 0.2°C.
* If baby's temperature is less than 36.3°C on 1 measurement, the isolette set temperature will be increased by 0.2°C.
* Once the baby's temperature is stable at greater than 36.7°C for 3 consecutive measurements 3 hours apart on an isolette set temp of 28.0°C, the baby will be transferred to an open crib. At this time, the baby will be dressed in one medium-weight sleeper with feet (or with socks if sleeper is footless), one hat, and a sleep sack. NO heavy blankets (such as bath blankets) or extra blankets are to be used.
* If the baby's temperature is less than 36.3°C on 1 measurement, they will be transferred back to the isolette and the weaning process will begin again.

Experimental Group: Conservative Wean

Weaning Process:

* If baby's temperature is greater than or equal to 37.2°C on 2 consecutive measurements 3 hours apart, the isolette set temperature will be lowered by 0.2°C.
* If baby's temperature is less than 36.3°C on 1 measurement, the isolette set temperature will be increased by 0.2°C.
* Once the baby's temperature is stable at greater than 37.2°C for 3 consecutive measurements 3 hours apart on an isolette set temp of 28.0°C, AND the baby is taking full caloric need feeds (at least 120 Kcal/kg/day), AND the baby is taking half of its feeds by mouth the baby will be transferred to an open crib. At this time, the baby will be dressed in one medium-weight sleeper with feet (or with socks if sleeper is footless), one hat, and a sleep sack. NO heavy blankets (such as bath blankets) or extra blankets are to be used.
* If the baby's temperature is stable at greater than 37.2°C for 4 consecutive measurements 3 hours apart on an isolette set temp of 28.0°C, or if the baby's temperature is greater than 37.9°C on an isolette set temp of 28.0°C, the baby will be transferred to an open crib regardless of feeding status. At this time, the baby will be dressed in one medium-weight sleeper with feet (or with socks if sleeper is footless), one hat, and a sleep sack. NO heavy blankets (such as bath blankets) or extra blankets are to be used.
* If the baby's temperature is less than 36.3 degrees Celsius on 1 measurement, they will be transferred back to the isolette and the weaning process will begin again.

Research Significance and Future Research:

This study will provide data regarding the weaning of thermoregulatory support in preterm infants, and could have significant economic impact for the university if there is a significant difference in length of stay between the study groups. Future research will focus on long-term effects on outcomes such as nutritional status in infancy and BMI in childhood if neonates do require greater caloric intake if they are weaned from thermoregulatory support faster.

Bibliography:

1. Dollberg S, Mimouni FB, Weintraub V. (2004) Energy expenditure in infants weaned from a convective incubator. American Journal of Perinatology. 21(5):253-6
2. Hackman P. (2001) Recognizing and understanding the cold-stressed term infant. The Journal of Neonatal Nursing. 20(8):35-41
3. New K, Flenady V, Davies MW. (2007) Transfer of preterm infants from incubator to open cot at lower versus higher body weight. The Cochrane Database of Systematic Reviews. 4.
4. Sherman TI, Greenspan JS, St. Clair N, Touch S, Shaffer T. (2006) Optimizing the neonatal thermal environment. Neonatal Network; The Journal of Neonatal Nursing. 25(4):251-60
5. Short MA. (1998) A comparison of temperature in VLBW infants swaddled versus unswaddled in a double-walled incubator in skin control mode. Neonatal Network; The Journal of Neonatal Nursing. 17(3):25-31
6. Weintraub V, Mimouni FB, Dollberg S. (2007) Changes in energy expenditure in preterm infants during weaning: A randomized comparison of two weaning methods from an incubator. Pediatric Research. 61(3):341-4

ELIGIBILITY:
Inclusion Criteria:

* Live born preterm infants from 26 and 0/7 weeks gestation to 34 and 6/7 weeks gestation
* Require thermoregulatory support
* Are able to take feeds
* Are presumed to be able to take oral feeds in the future

Exclusion Criteria:

* Preterm infants less than 26 and 0/7 weeks gestation
* Preterm infants greater than 34 and 6/7 weeks gestation
* Infants that do not require thermoregulatory support
* Infants that will not be able to have enteral feeds
* Infants with endocrine disease
* Infants with congenital anomalies
* Infants with grade 3 or 4 intraventricular hemorrhage or other severe neurologic disability
* Infants requiring long-term sedation
* Infants that die within 7 days of birth

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-10-22 (Actual); Primary Completion 2011-01-26 (Actual); Study Completion 2011-01-26 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | Hospital discharge

SECONDARY OUTCOMES:
Weight gain | When patient is on 120 cal/kg/day dietary intake
Caloric requirement | When patient is changed to oral ad lib demand feeds

CONTACTS AND LOCATIONS:
Overall Officials: Sarah B Patton, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- Columbia Regional Hospital, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No